CLINICAL TRIAL: NCT05417828
Title: Robotic Rehabilitation for Stroke Survivors
Status: Not yet recruiting | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Department of Neurology Jacobs School of Medicine and Biomedical Sciences University at Buffalo. (Unknown)
Responsible Party: Principal Investigator, Amit Kandel, MD, MBA, Principal Investigator, State University of New York at Buffalo
Other Study IDs: STUDY00005946
Record Dates: First submitted 2022-06-05; First posted 2022-06-14 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Chronic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participant with Chronic stroke: 1. Participants over 18 years of age
  2. Participants should be able to understand the verbal cues during the training
  Interventions: Device: Emulation of Active Daily Living tasks with a robotic device (SPINDLE)

INTERVENTIONS:
Device: Emulation of Active Daily Living tasks with a robotic device (SPINDLE) — SPINDLE will provide an assistive and resistive force to aid in rehabilitating the subject's upper limb

SUMMARY:
Pilot study on the physiological response of robotic rehabilitation therapy for improving the performance of activities of daily living of stroke patients

DETAILED DESCRIPTION:
The purpose of this research is to study the feasibility of the robotic therapy that can train activities of daily living tasks for chronic stroke patients. The participant will be involved in a feasibility study (one-time visit) to prove the efficacy of the robotic device with different force feedback (assistive and resistive force) and other feedback such as VR (virtual reality). We will collect movement data from a motion capture system and sEMG sensors that measure muscle activity to monitor the effect of a robotic rehabilitation device, named Spherical Parallel Instrument for Daily Living Emulation (SPINDLE). We will use a robotic therapy device to practice activities during daily living. This pilot study will be used to understand the effect of SPINDLE to translate the device as a home-based training for chronic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults with chronic stroke, which affected their upper limb motor functions
* Adults could able to understand the verbal cues during the training

Exclusion Criteria:

* Adults with chronic stroke, who did not lose their upper limb motor functions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study participant needs to have minimal strength to move the robot. The participant needs to be able to understand the instructions during the experiment.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-05 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
Kinematic change of the upper limb during ADLs | immediately after the intervention
  The max and range of motion of shoulder, elbow, and wrist joint for each task
Score of activities of daily living(ADL) tasks | immediately after the intervention
  We will use ARM-ULA standard score sheet to measure the performance of ADLs
Muscle activation change of the upper limb during ADLs | immediately after the intervention
  The subject will be asked to perform activities of daily living tasks with the passive SPINDLE. Upper limb range of motion and muscle activation will be quantified.

SECONDARY OUTCOMES:
Usability measure | immediately after the intervention
  Questionnaire will be provided to the user to obtain qualitative feedback

CONTACTS AND LOCATIONS:
Overall Officials: Jiyeon Kang, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, North Campus, Furnas 809, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data will be shared upon request to PI.
Time Frame: After the study is completed
Access Criteria: The personnel who is requesting the data needs to explain how the data will be used in their research.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT05417828/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT05417828/ICF_001.pdf